CLINICAL TRIAL: NCT02306889
Title: An Open Label, Balanced, Randomized, Two-treatment, Two -Period, Two -Sequence, Crossover Bioequivalence Study Comparing a Single Oral Dose of Fenofibrate 130 mg Capsules of Ohm Laboratories Inc. USA (a Subsidiary of Ranbaxy Pharmaceutical Inc.) With Antara® 130 mg Capsules (Containing Fenofibrate 130 mg) of Oscient Pharmaceuticals Corporation USA, in Healthy, Adult, Male, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Fenofibrate Capsules, 130 mg Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 102_FENOF_10
Record Dates: First submitted 2014-11-24; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Fenofibrate Capsules, USP 130 mg
  Interventions: Drug: Fenofibrate
- Reference (Active Comparator): ANTARA® (fenofibrate) Capsules 130 mg
  Interventions: Drug: ANTARA® (fenofibrate)

INTERVENTIONS:
Drug: Fenofibrate — 130mg Capsules
  Arms: Test
Drug: ANTARA® (fenofibrate) — 130mg Capsules
  Arms: Reference

SUMMARY:
The study was conducted as an open label, balanced, randomized, two-treatment, two-period, two-sequence, crossover bioequivalence study comparing a single oral dose of fenofibrate capsules, USP 130 mg, of Ohm Laboratories Inc. USA (a subsidiary of Ranbaxy Pharmaceutical Inc.) with Antara® (fenofibrate) Capsules 130 mg of Oscient Pharmaceuticals Corporation USA, in healthy, adult, male, human subjects under fasting condition.

DETAILED DESCRIPTION:
The subjects were subjected to breath test for alcohol and test for drugs of abuse (opioids and cannabinoids) in urine prior to admission in each period.

All subjects fasted overnight for at least 10 hours before the morning dose and for 4 hours post-dose during each period of the study. A single oral dose of either test (T) or reference (R) was administered with 240 mL of drinking water at ambient temperature under supervision of trained study personnel. Both test and reference products were administered to all the study subjects, one in each period (except subject numbers 17, 27 and 42).

Blood samples were collected at Predose (duplicate) and at 1.000, 2.000, 2.500, 3.000, 3.500, 4.000, 4.500, 5.000, 5.500, 6.000, 6.500, 7.000, 7.500, 8.000, 8.500, 9.000, 10.000, 11.000, 12.000, 16.000, 24.000, 36.000, 48.000, 72.000 and 96.000 hours post dose, in pre-chilled vacutainers, under low light condition, in each period from all completed subjects. The pre-dose blood samples in each period were collected in duplicate (2 x 5 mL), within a period of 1.5 hour before dosing.

The actual end time of collection of each blood sample was recorded. During the course of the study, safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis at screening). Adverse event monitoring was done throughout the study. Laboratory parameters of hematology and biochemistry were repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Volunteers who met the following criteria were included in the study

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for his/her height as per the Life Insurance Corporation of India height/weight chart for non-medical cases
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* History of hypersensitivity to fenofibrate or any other related drug.
* Subjects with history of hepatic or severe renal dysfunction, including primary biliary cirrhosis.
* Subjects with history of unexplained persistent liver function abnormality.
* Subject had history of myalgia, muscle tenderness or weakness or myopathy.
* History of abdominal pain in one week preceding the study.
* History of recurrent headache and/or back pain.
* History of constipation and/or nausea in one week preceding the study.
* History and/or any finding of gall bladder disease.
* History of pancreatitis.
* History of drug-induced rash and/or pruritis. - Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Subject had laboratory test parameter(s), which is/are outside acceptable limits and is judged clinically significant.
* Subject had history of serious medical illnesses including but not limited to gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes, glaucoma, any serious, potentially life-threatening illness.
* Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that might impair the ability to provide, written informed consent.
* Subject was a regular smoker, who smoked more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* Subject had history of drug dependence or excessive alcohol intake on a habitual basis or has difficulty in abstaining for the duration of each study period or has consumed alcohol 48 hours prior to admission.
* Subject had used an enzyme modifying drugs within 30 days prior to admission of this study.
* Subject had participated in a clinical trial within 12 weeks preceding admission of this study (except for subjects who dropout / are withdrawn from the previous study prior to period 1 dosing)
* Subject had donated and/or lost more than 350 mL of blood in the past 3 months, including blood loss in this study.
* Consumption of alcohol for 48 hours prior to admission.
* Subject had problem(s) in complying with the study protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of fenofibric acid | 0-96 hrs
Peak Plasma Concentration (Cmax) of fenofibric acid | 0-96 hrs

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm